CLINICAL TRIAL: NCT02527434
Title: A Phase II, Multi-Center, Open-Label Study of Tremelimumab Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Study of Tremelimumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4884C00001; 2015-002934-32 (EudraCT Number)
Record Dates: First submitted 2015-08-12; First posted 2015-08-19 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Urothelial Bladder Cancer; Triple-negative Breast Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Urothelial bladder cancer, Triple-negative breast cancer, Pancreatic ductal adenocarcinoma, Advanced Solid Tumors, Tremelimumab, MEDI4736, ORR
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- treme mono to be sequenced to MEDI4736 mono or combination (Experimental): tremelimumab monotherapy, with the option for eligible patients to be sequenced to MEDI4736 monotherapy or MEDI4736 + tremelimumab combination therapy after progressive disease (PD)
  Interventions: Biological: Tremelimumab monotherapy; Biological: MEDI4736 monotherapy; Biological: MEDI4736 + tremelimumab combination therapy

INTERVENTIONS:
Biological: Tremelimumab monotherapy — IV infusion
Biological: MEDI4736 monotherapy — IV infusion
Biological: MEDI4736 + tremelimumab combination therapy — IV infusion

SUMMARY:
A Phase II, Multi-Center, Open-Label Study of Tremelimumab Monotherapy in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is an open-label, multi-center study to determine the efficacy and safety of tremelimumab in the treatment of different cohorts of patients with selected advanced solid tumors. If eligible and at the discretion of the Investigator, after confirmed disease progression on tremelimumab monotherapy or during follow-up, patients will have the option of being sequenced to MEDI4736 (MedImmune 4736) monotherapy or MEDI4736 + tremelimumab combination therapy, for up to 12 months or until disease progression, whichever comes sooner.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically documented solid tumor malignancies, including but not limited to 1 of the following: UBC, Metastatic PDAC, TNBC; Are intolerant, are ineligible for, or have refused treatment with standard first-line therapy; 2. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) (preferred) or magnetic resonance imaging (MRI) scans and that is suitable for accurate repeated measurements.

Exclusion criteria:

1. Any concurrent chemotherapy, biologic, or hormonal therapy for cancer Treatment; 2. History of leptomeningeal carcinomatosis; 3. Active or prior documented autoimmune or inflammatory disorders; 4. Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 14 days prior to study treatment start; 5. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms; 6. Known allergy or hypersensitivity to IP or any IP excipient

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharma Padmanee, MD, PhD, Principal Investigator — Anderson Cancer Center, the University of Texas
Locations (12):
- United States (3):
  - Research Site, San Francisco, California
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Wilrijk
- Netherlands (2):
  - Research Site, Groningen
  - Research Site, Utrecht
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Lodz
- South Korea (2):
  - Research Site, Daejeon
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3801&filename=D4884C00001-statistical-analysis-plan-edition-2_%2022Jun2018_Published%20on%20CARA-redact.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3801&filename=D4884C00001-csp-v4_final_clean_13Sep2018-redact.pdf
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4884C00001&attachmentIdentifier=e176d601-e473-4d9e-b20b-051d9448cee1&fileName=d4884c00001-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 patients with select advanced solid tumors were treated in this phase II, open-label, multi-center study from November 2015. Primary data cut off date: 17 February 2018. Final data cut off date: 31 December 2018.
Pre-assignment Details: The patients were split into 3 different analysis cohorts based on their tumor types: urothelial bladder cancer (UBC), triple-negative breast cancer (TNBC) and pancreatic ductal adenocarcinoma (PDAC).
Groups:
- UBC Cohort: Patients with UBC entered the initial tremelimumab monotherapy phase and were administered tremelimumab via intravenous (IV) infusion at a dose of 750 milligrams (mg) once every 4 weeks (q4w) for 7 doses (cycles), then every 12 weeks (q12w) for 2 additional cycles, for up to a total of 12 months or until confirmed progressive disease (PD).
  Eligible patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were given the option for retreatment with tremelimumab monotherapy or to be sequenced to receive MEDI4736 (durvalumab) + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months or to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
- TNBC Cohort: Patients with TNBC entered the initial tremelimumab monotherapy phase and were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
  Eligible patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were given the option for retreatment with tremelimumab monotherapy or to be sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months or to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
- PDAC Cohort: Patients with PDAC entered the initial tremelimumab monotherapy phase and were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
  Eligible patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were given the option for retreatment with tremelimumab monotherapy or to be sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months or to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
Period: Overall Study
Arm/Group | UBC Cohort | TNBC Cohort | PDAC Cohort
Started (Full Analysis Set (FAS)) | 32 | 12 | 20
Started Retreatment Phase (COMBO) (COMBO Analysis Set) | 7 | 5 | 4
Started Retreatment Phase (MEDI) (MEDI Analysis Set) | 4 | 0 | 1
Completed | 4 | 1 | 0
Not Completed | 28 | 11 | 20
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Death | 19 | 6 | 17
Not completed — Withdrawal by Subject | 5 | 3 | 3
Not completed — Reason Not Specified | 1 | 0 | 0
Not completed — Site closure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Groups:
- UBC Cohort: Patients with UBC entered the initial tremelimumab monotherapy phase and were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
  Eligible patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were given the option for retreatment with tremelimumab monotherapy or to be sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months or to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
- Total: Total of all reporting groups
Arm/Group | UBC Cohort | TNBC Cohort | PDAC Cohort | Total
Number analyzed (Participants) | 32 | 12 | 20 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 8 | 14 | 35
  >=65 years | 19 | 4 | 6 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 9 | 27
  Male | 26 | 0 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 31 | 12 | 20 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 11 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 21 | 1 | 8 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Confirmed Overall Response During Tremelimumab Monotherapy Phase
Description: Objective response rate (ORR) during the initial tremelimumab monotherapy phase was assessed by the site Investigator using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) and was defined as the percentage of patients with a confirmed overall response of complete response (CR) or partial response (PR) and was based on all treated patients who had measurable disease at baseline (Day 1). 95% confidence intervals (CIs) were calculated using the Clopper Pearson method.
Time Frame: From baseline to 12 months in the tremelimumab monotherapy phase
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- UBC - Tremelimumab Monotherapy: Patients with UBC were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
- TNBC - Tremelimumab Monotherapy: Patients with TNBC were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
- PDAC - Tremelimumab Monotherapy: Patients with PDAC were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Percentage of Patients | 18.8 [7.2 to 36.4] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 16.8]

2. Secondary Outcome: Median Duration of Response (DoR) During Tremelimumab Monotherapy Phase
Description: DoR during the initial tremelimumab monotherapy phase was assessed by the site Investigator using RECIST 1.1 and was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The time of the initial response was defined as the latest of the dates contributing toward the first visit response of CR or PR. If a patient did not progress following a response, then their DoR was censored at the progression-free survival (PFS) censoring time. DoR was not defined for those patients who did not have documented response. Median DoR was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to 12 months in the tremelimumab monotherapy phase
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Months | NA [NA to NA] — DoR was not estimable in this cohort | 12.9 [12.9 to 12.9] | NA [NA to NA] — DoR was not estimable in this cohort

3. Secondary Outcome: Disease Control Rate (DCR) During Tremelimumab Monotherapy Phase
Description: DCR during the initial tremelimumab monotherapy phase was defined as the percentage of patients who had a best objective response (BoR) of CR or PR in the first 3 months (PDAC patients) or 4 months (UBC and TNBC patients) and 12 months (all patients), or who had demonstrated stable disease (SD) for a minimum interval of 3, 4 or 12 months following the start of study treatment. DCR was determined programmatically based on RECIST 1.1 using site Investigator data and all data up until the first progression event. 95% CIs were calculated using the Clopper Pearson method.
Time Frame: From baseline to 12 months in the tremelimumab monotherapy phase
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Percentage of patients
  DCR at 3 or 4 months | 25.0 [11.46 to 43.40] | 8.3 [0.21 to 38.48] | 0.0 [0.00 to 16.84]
  DCR at 12 months | 21.9 [9.28 to 39.97] | 8.3 [0.21 to 38.48] | 0.0 [0.00 to 16.84]

4. Secondary Outcome: Median PFS During Tremelimumab Monotherapy Phase
Description: PFS during the initial tremelimumab monotherapy phase was assessed by the site Investigator using RECIST 1.1 and was defined as the time from the date of enrollment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from therapy or received another anticancer therapy prior to progression. Progression events that did not occur within 3 months (PDAC patients) or 4 months (UBC/TNBC patients) of the last evaluable assessment (or first dose) were censored. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to 12 months in the tremelimumab monotherapy phase
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Months | 2.63 [1.77 to NA] — The upper limit was not estimable in this cohort. | 3.58 [1.40 to 4.04] | 1.77 [1.38 to 2.92]

5. Secondary Outcome: Best Objective Response (BoR) During Tremelimumab Monotherapy Phase
Description: BoR during the initial tremelimumab monotherapy phase was calculated based on the overall visit responses from each RECIST 1.1 assessment and was defined as the best response a patient had during their time in the study (from CR, PR, SD, PD or not evaluable [NE]) obtained among all tumor assessment visits from baseline until end of treatment or determination of PD. The BoR was summarized by percentage of patients for each category (CR, PR, SD, PD, and NE).
Time Frame: From baseline to 12 months in the tremelimumab monotherapy phase
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Number; unit: Percentage of Patients
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Percentage of Patients
  CR | 6.3 | 0.0 | 0.0
  PR | 12.5 | 8.3 | 0.0
  SD | 9.4 | 0.0 | 0.0
  PD | 68.8 | 91.7 | 90.0
  NE | 3.1 | 0.0 | 10.0

6. Secondary Outcome: Median Overall Survival (OS) During Tremelimumab Monotherapy Phase
Description: OS was defined as the time from the date of first dose until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. OS is presented from start of tremelimumab monotherapy phase and includes the retreatment phase if the patient entered the corresponding treatment phase.
  Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to final data cut-off date
Population: Analysis was performed on the FAS (all treated patients who received at least 1 dose of tremelimumab monotherapy).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | UBC - Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC - Tremelimumab Monotherapy
Number analyzed (Participants) | 32 | 12 | 20
Months | 10.32 [5.91 to 24.61] | 12.88 [2.53 to NA] — Upper limit was not estimable in this cohort. | 3.98 [2.83 to 5.13]

7. Secondary Outcome: Percentage of Patients With Confirmed Overall Response During Retreatment Phase
Description: ORR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR and was based on all treated patients who had measurable disease at baseline (Day 1) and who sequenced to durvalumab monotherapy (MEDI treatment phase) or durvalumab + tremelimumab combination therapy (COMBO treatment phase). 95% CIs were calculated using the Clopper Pearson method.
Time Frame: From baseline to 12 months in retreatment phase
Population: Analysis was performed on the MEDI and COMBO analysis sets (all patients who were treated with tremelimumab, received at least 1 dose of durvalumab monotherapy or durvalumab + tremelimumab combination therapy as applicable, and who had a baseline tumor assessment prior to dosing).
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Groups:
- UBC - COMBO: Eligible UBC patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months.
- TNBC - COMBO: Eligible TNBC patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months.
- PDAC - COMBO: Eligible PDAC patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were sequenced to receive durvalumab + tremelimumab combination therapy (also referred to as COMBO; durvalumab 1.5 g via IV infusion q4w in combination with tremelimumab 75 mg via IV infusion q4w for up to 4 cycles each, followed by durvalumab 1.5 g via IV infusion q4w) for up to a total of 8 months.
- UBC- MEDI: Eligible UBC patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were sequenced to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
- PDAC - MEDI: Eligible PDAC patients with confirmed PD on tremelimumab monotherapy or during the follow-up period were sequenced to receive durvalumab monotherapy (also referred to as MEDI; 1.5 g via IV infusion q4w) for up to a total of 12 months.
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Percentage of Patients | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2] | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 97.5]

8. Secondary Outcome: Median DoR During Retreatment Phase
Description: DoR during the retreatment phase was assessed by the site Investigator using RECIST 1.1 and was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The time of the initial response was defined as the latest of the dates contributing toward the first visit response of CR or PR. If a patient did not progress following a response, then their DoR was censored at the PFS censoring time. DoR was not defined for those patients who did not have documented response. Median DoR was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to 12 months in retreatment phase
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Months | NA [NA to NA] — No DoR data were available for this cohort. | NA [NA to NA] — No DoR data were available for this cohort. | NA [NA to NA] — No DoR data were available for this cohort. | 7.3 [7.3 to 7.3] | NA [NA to NA] — DoR was not estimable in this cohort

9. Secondary Outcome: DCR During Retreatment Phase
Description: DCR during the retreatment phase was defined as the percentage of patients who had a BoR of CR or PR in the first 3 months (PDAC patients) or 4 months (UBC and TNBC patients) or who had demonstrated SD for a minimum interval of 3 or 4 months following the start of study treatment. DCR was determined programmatically based on RECIST 1.1 using site Investigator data and all data up until the first progression event. 95% CIs were calculated using the Clopper Pearson method.
Time Frame: From baseline to 4 months in retreatment phase
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Percentage of Patients | 28.6 [3.67 to 70.96] | 20.0 [0.51 to 71.64] | 25.0 [0.63 to 80.59] | 25.0 [0.63 to 80.59] | 0.0 [0.00 to 97.50]

10. Secondary Outcome: Median PFS During Retreatment Phase
Description: PFS during the retreatment phase was assessed by the site Investigator using RECIST 1.1 and defined as the time from the date of enrollment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from therapy or received another anticancer therapy prior to progression.
  Progression events that did not occur within 3 months (PDAC patients) or 4 months (UBC/TNBC patients) of the last evaluable assessment (or first dose) were censored. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to 12 months in retreatment phase
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Months | 2.83 [1.81 to 3.65] | 0.99 [0.92 to NA] — Upper limit was not estimable in this cohort. | 2.86 [1.87 to 3.52] | 2.86 [1.81 to 6.62] | 1.84 [1.84 to 1.84]

11. Secondary Outcome: BoR During Retreatment Phase
Description: BoR during the retreatment phase was calculated based on the overall visit responses from each RECIST 1.1 assessment and was defined as the best response a patient had during their time in the study (from CR, PR, SD, PD or NE) obtained among all tumor assessment visits from baseline until end of treatment or determination of PD. The BoR was summarized by percentage of patients for each category (CR, PR, SD, PD, and NE).
Time Frame: From baseline to 12 months in retreatment phase
Population: as for outcome 7
Measure: Number; unit: Percentage of Patients
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Percentage of Patients
  CR | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  PR | 0.0 | 0.0 | 0.0 | 25.0 | 0.0
  SD | 14.3 | 20.0 | 0.0 | 0.0 | 0.0
  PD | 71.4 | 80.0 | 100.0 | 75.0 | 100.0
  NE | 14.3 | 0.0 | 0.0 | 0.0 | 0.0

12. Secondary Outcome: Median OS During Retreatment Phase
Description: OS during the retreatment phase was defined as the time from the date of first dose until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline in retreatment phase to final data cut-off date
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 1
Months | 11.86 [5.91 to NA] — Median and upper limit was not estimable in this cohort. | 33.05 [9.69 to 33.05] | 7.18 [3.98 to 18.76] | 16.53 [7.56 to 32.39] | 4.14 [NA to NA] — Lower and upper limits were not estimable in this cohort.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 (i.e. first dose) up until 90 days following the end of treatment in the tremelimumab monotherapy phase and the retreatment phase (up to a total of 15 months per treatment phase).
Groups:
- UBC- Tremelimumab Monotherapy: Patients with UBC were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
- PDAC- Tremelimumab Monotherapy: Patients with PDAC were administered tremelimumab via IV infusion at a dose of 750 mg q4w for 7 cycles, then q12w for 2 additional cycles, for up to a total of 12 months or until confirmed PD.
Arm/Group | UBC- Tremelimumab Monotherapy | TNBC - Tremelimumab Monotherapy | PDAC- Tremelimumab Monotherapy | UBC - COMBO | TNBC - COMBO | PDAC - COMBO | UBC- MEDI | PDAC - MEDI
All-Cause Mortality (participants affected / at risk) | 13/32 | 4/12 | 12/20 | 4/7 | 2/5 | 4/4 | 4/4 | 1/1
Serious Adverse Events (participants affected / at risk) | 18/32 | 4/12 | 11/20 | 3/7 | 2/5 | 3/4 | 1/4 | 0/1
Other Adverse Events (participants affected / at risk) | 30/32 | 10/12 | 19/20 | 7/7 | 5/5 | 4/4 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UBC- Tremelimumab Monotherapy (N=32) | TNBC - Tremelimumab Monotherapy (N=12) | PDAC- Tremelimumab Monotherapy (N=20) | UBC - COMBO (N=7) | TNBC - COMBO (N=5) | PDAC - COMBO (N=4) | UBC- MEDI (N=4) | PDAC - MEDI (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UBC- Tremelimumab Monotherapy (N=32) | TNBC - Tremelimumab Monotherapy (N=12) | PDAC- Tremelimumab Monotherapy (N=20) | UBC - COMBO (N=7) | TNBC - COMBO (N=5) | PDAC - COMBO (N=4) | UBC- MEDI (N=4) | PDAC - MEDI (N=1)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 2 (3) | 4 (7) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (20) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (3) | 2 (2) | 2 (3) | 1 (5) | 1 (1) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 2 (2) | 5 (5) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (5) | 7 (7) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular fragility (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any or all of the results of the Research by the PI requires prior written consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT02527434/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02527434/SAP_000.pdf